CLINICAL TRIAL: NCT02887001
Title: Impact of Clinical Pharmacist on the Quality and Cost of the Therapeutic Management of Patients in Two Medical Services of a Teaching Hospital
Acronym: ImpactPharma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LOCAL/2010/JMK-01; 2010-A00186-35 (Other: ANSM)
Record Dates: First submitted 2016-08-24; First posted 2016-09-01 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2016-07

CONDITIONS: Admitted to Infectiology or Internal Medicine Wards
Keywords: cost study; clinical pharmacist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMO (Other)
  Interventions: Other: Pharmacist consultation

INTERVENTIONS:
Other: Pharmacist consultation

SUMMARY:
Incomplete information or poorly communicated to the transitional stages of the patient's drug therapy hospitalized cause medication errors. These steps are the admission, transfer within the institution and hospital discharge to home or another institution.

The adequacy of the prescription recommendations of good practice is not always optimal.

The cost of taking drug therapy and iatrogenic risks preventable drug-related weighs more and more heavily in health spending and in the prolongation of hospitalization or re hospitalization.

Clinical pharmacy widely practiced in the Anglo-Saxon countries has demonstrated its effectiveness on these three themes; it seems appropriate to assess this practice in the environment of the French health system.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted in in infectious and tropical diseases unit or the internal medicine unit

Exclusion Criteria:

* none

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07-01 (Actual); Study Completion 2012-07-01 (Actual)

PRIMARY OUTCOMES:
Number of prescriptions | 11 weeks

REFERENCES:
- [Result] Leguelinel-Blache G, Dubois F, Bouvet S, Roux-Marson C, Arnaud F, Castelli C, Ray V, Kinowski JM, Sotto A. Improving Patient's Primary Medication Adherence: The Value of Pharmaceutical Counseling. Medicine (Baltimore). 2015 Oct;94(41):e1805. doi: 10.1097/MD.0000000000001805. PMID 26469927